CLINICAL TRIAL: NCT04827927
Title: The Effect of Closed-Loop Versus Conventional Ventilation on Mechanical Power - a Multicenter Crossover Randomized Clinical Trial
Brief Title: The Effect of Closed-Loop Versus Conventional Ventilation on Mechanical Power
Acronym: INTELLiPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Reinier de Graaf Groep (Other); Dijklander Ziekenhuis (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr. Marcus J. Schultz, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INTELLiPOWER
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Mechanical Ventilation; Mechanical Power

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTELLiVENT-ASV (Experimental): Use of INTELLiVENT-ASV during 3 hours with 30 minutes wash-out time before.
  Interventions: Procedure: Procedure: INTELLiVENT-ASV
- Conventional Ventilation (Active Comparator): Use of conventional ventilation during 3 hours with 30 minutes wash-out time before.
  Interventions: Procedure: Procedure: Conventional ventilation

INTERVENTIONS:
Procedure: Procedure: INTELLiVENT-ASV — With INTELLiVENT-ASV, the patient's conditions, 'ARDS', 'Chronic Hypercapnia' or 'Traumatic Brain Injury' can be chosen, if applicable. The controllers for minute volume, PEEP and FiO2 are all activated, and the target shifts for etCO2 and SpO2 are adjusted, if necessary.
  Arms: INTELLiVENT-ASV
Procedure: Procedure: Conventional ventilation — With conventional ventilation, the same etCO2 and SpO2 levels are targeted as with INTELLiVENT-ASV, but here the caregiver is fully responsible for choosing the settings.
  Arms: Conventional Ventilation

SUMMARY:
Several studies suggest fully-automated ventilation to ventilate with a lower amount of MP in unselected ICU patients, patients after cardiac surgery, and patients with and without ARDS. The current study will directly compare the amount of MP in invasively ventilated critically ill patients by calculating MP breath-by-breath, using the various equations proposed in the literature.

DETAILED DESCRIPTION:
Rationale:

Mechanical ventilation can cause ventilator-induced lung injury (VILI). Lung protective ventilation, consisting of a low tidal volume (VT), a low plateau pressure (Pplateau) and a low driving pressure (ΔP) improves survival and shortens duration of ventilation in patients with acute respiratory distress syndrome (ARDS). Lung protective ventilation may also benefit critically ill patients with respiratory failure not caused by ARDS. 'Mechanical Power of ventilation' (MP), the amount of energy per time transferred from the ventilator to the respiratory system, is a summary variable that includes all the components that play a role in VILI. With fully-automated closed-loop ventilation, these components are no longer set by the operator, but under control of the algorithms in the ventilator.

Objective:

To compare MP under INTELLiVENT-adaptive support ventilation (ASV), a fully-automated closed-loop ventilation, with MP under conventional ventilation.

Hypothesis:

INTELLiVENT-ASV compared to conventional ventilation results in a lower MP.

Study design:

National, multicenter, crossover, randomized clinical trial.

Study population:

Invasively ventilated critically ill patients.

Methods:

The ventilator will be randomly switched between INTELLiVENT-ASV for 3 hours and conventional ventilation for 3 hours. The amount of MP is calculated using various equations proposed in the literature.

Study endpoints:

The primary endpoint is the amount of MP with each form of invasive ventilation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Differences in burden and risks of the two ventilation strategies compared in the current study are not expected. Both modes of ventilation are interchangeably used as part of standard care in the participating centers. No other interventions are performed. Neither the collection of demographic and outcome data, nor the capturing of ventilation characteristics causes harm to patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to one of the participating ICUs;
* Receiving invasive ventilation through a standard endotracheal (i.e., oral) tube;
* Expected to be ventilated > 24 hours; and
* Ventilation is applied by a ventilator that can provide INTELLiVENT-ASV and conventional ventilation.

Exclusion Criteria:

* Age under 18 years;
* No written informed consent;
* Morbidly obese; and
* Any contra-indication for use of INTELLiVENT-ASV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The amount of MP delivered with each form of invasive ventilation | 3 hours per ventilation mode
  The amount of MP delivered with INTELLiVENT-ASV and conventional ventilation

SECONDARY OUTCOMES:
Duration of ventilation | first 28 days after start of ventilation
  Duration of ventilation in survivors
ICU-length and hospital of stay | first 28 days after start of ventilation
  Length of stay in the intensive care unit and in the hospital
28 day-mortality | first 28 days after start of ventilation
  Any death during ICU-, hospital-stay and within 28 days
Tidal volume | 3 hours per ventilation mode
  Tidal volume in ml/kg
Respiratory rate | 3 hours per ventilation mode
  Respiratory rate per minute
Pmax | 3 hours per ventilation mode
  Maximum airway pressure in cmH2O
Driving pressure | 3 hours per ventilation mode
  Difference between end-inspiratory pressure and total Positieve End Expiratory Pressure in cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD, PhD, Principal Investigator — Department of Intensive Care, Amsterdam University Medical Centre - location AMC; Frederique Paulus, PhD, Study Director — Department of Intensive Care, Amsterdam University Medical Centre - location AMC; Laura A Buiteman-Kruizinga, RN, BSc, Study Director — Department of Intensive Care, Amsterdam University Medical Centre - location AMC
Locations (3):
- Netherlands (3):
  - Academic Medical Center, Amsterdam, North Holland
  - Reinier de Graaf Gasthuis, Delft
  - Dijklander Ziekenhuis, Hoorn

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buiteman-Kruizinga LA, Serpa Neto A, Botta M, List SS, de Boer BH, van Velzen P, Buhler PK, Wendel Garcia PD, Schultz MJ, van der Heiden PLJ, Paulus F; INTELLiPOWER-investigators. Effect of automated versus conventional ventilation on mechanical power of ventilation-A randomized crossover clinical trial. PLoS One. 2024 Jul 30;19(7):e0307155. doi: 10.1371/journal.pone.0307155. eCollection 2024. PMID 39078857

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT04827927/Prot_SAP_000.pdf